CLINICAL TRIAL: NCT01995487
Title: BioNIR Ridaforolimus Eluting Coronary Stent System (BioNIR) In Coronary Stenosis Trial
Brief Title: Study of BioNIR Drug Eluting Stent System in Coronary Stenosis
Acronym: BIONICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioNIR-001
Record Dates: First submitted 2013-11-12; First posted 2013-11-26 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Stenosis
Keywords: more comers; DES; BioNIR; ACS; non ACS; complex lesions
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: This is a Drug-Device combination Product.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioNIR (Experimental): The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0
  The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
  Interventions: Device: BioNIR
- Resolute (Active Comparator): The Endeavor Resolute Zotarolimus-Eluting Stent System consists of four subsystems:
  1. Endeavor Resolute Stent- a pre-mounted cobalt alloy based stent
  2. Delivery system (Rapid Exchange [RX] Coronary System)
  3. Polymer system
  4. Zotarolimus - drug The Resolute has a nominal drug dose of 1.6µg Zotarolimus per mm2 of the stent surface area.
  Interventions: Device: Resolute

INTERVENTIONS:
Device: BioNIR — drug-eluting stent
  Arms: BioNIR
Device: Resolute — drug-eluting stent
  Arms: Resolute

SUMMARY:
The BioNIR study aims to show that the BioNIR ridaforolimus eluting stent is non-inferior to the Resolute zotarolimus-eluting stent for the primary clinical endpoint of target lesion failure (TLF) at 12 months; that it is non-inferior to the Resolute for the secondary endpoint of angiographic in-stent late loss at 13 months; and that it is more cost-effective.

DETAILED DESCRIPTION:
The BioNIR is a prospective, multi-center, single-blind, two-arm, randomized clinical trial. The population will consist of subjects undergoing PCI for angina (stable or unstable), silent ischemia, NSTEMI, and recent STEMI. Complex lesions are allowed. There is no limit to the number of lesions per vessel or individual lesion length; however, the total planned stenting in the coronary tree cannot exceed 100mm.

Randomization will be stratified by the presence of medically treated diabetes vs. no medically treated diabetes, acute coronary syndrome (ACS) vs. non-ACS, and by site. Lesions planned to be treated must be declared and recorded at time of randomization. Planned staged procedures, if necessary, must be declared immediately post procedure.

Clinical follow-up will be performed at 30 days, 6 months, and 1, 2, 3, 4, and 5 years post randomization. 200 patients at participating North American sites will be consented for planned angiographic follow-up at 13 months after enrollment, with 100 of these patients consented to undergo planned IVUS at baseline and at 13 months following randomization.

The primary endpoint is Target Lesion Failure (TLF) at 12 months, defined as the composite of cardiac death, target vessel-related myocardial infarction, or ischemia-driven target lesion revascularization.

Clinical Secondary Endpoints to be evaluated at 30 days, 6 months, and 1, 2, 3, 4 and 5, except as noted:

* Device, Lesion, and Procedure Success at time of baseline procedure
* TLF at 30 days, 6 months, and 2, 3, 4 and 5 years defined as the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR.
* Major adverse cardiac events (MACE; the composite rate of cardiac death, any MI or ischemia-driven TLR)
* Target vessel failure (TVF; the composite rate of death, target vessel related MI or ischemia-driven TVR)
* All-cause mortality
* Cardiac death
* Myocardial Infarction
* Target Vessel Related MI
* Ischemia-driven TLR
* Ischemia-driven TVR
* Stent Thrombosis (ARC definite and probable)

Angiographic Sub-Study Secondary Endpoint to be evaluated at 13 months:

• Angiographic in-stent and in-segment late loss

IVUS Sub-Study Secondary Endpoint to be evaluated at 13 months:

* In-stent percent neointimal hyperplasia
* Stent mal-apposition

A key component of this trial will be a prospective assessment of health care resource utilization, costs and cost effectiveness. A separate cost effectiveness assessment plan describes the data collection and analysis.

Sample Size Consideration: From recent US trials of best in class DES (Xience V, Promus Element and Resolute), the 1-year TLF rate in patients with non-complex lesions not undergoing routine angiographic follow-up is approximately 3.8%. Using the assumption of the more-comers' design, the 1-year event rate will be conservatively increased by 50% (assuming enrollment rate for complex patients/lesions is 50% with double the standard event rate) - thus 5.8%. Therefore, with a one-sided 95% upper bound of the confidence interval of 3.3% (a relative 57% margin) and 1:1 randomization, enrolling 1810 patients (905 per group) provides 90% power to demonstrate non-inferiority. Assuming 95% follow-up rate at 1 year, approximately 1906 patients will be enrolled (953 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for PCI including angina/silent ischemia/NSTEMI/recent STEMI
* Non-target vessel PCI allowed prior to randomization depending on time interval and certain conditions
* Patient/legal guardian willing & able to provide informed written consent & comply with follow-up visits & testing schedule
* Target lesion(s) must be located in native coronary artery/bypass graft conduit w/visually estimated diameter ≥2.5mm to ≤4.25mm.
* Complex lesions allowed, including calcified, presence of thrombus, CTO, bifurcation (except as per exclusion criteria #30), ostial RCA, tortuous, bare metal stent restenotic, protected left main, and saphenous vein graft

Exclusion Criteria:

* STEMI within 24 hours of init. time of presentation to first treating hospital, or in whom enzyme levels (either CK-MB or Troponin) have not peaked
* PCI within 24 hours preceding baseline procedure
* Non-target lesion PCI in target vessel within 12 months of baseline procedure
* History of stent thrombosis
* Cardiogenic shock (persistent hypotension [systolic blood pressure <90mm/Hg for MT 30 min] or requiring pressors/hemodynamic support, including IABP)
* Subject is intubated
* Known LVEF <30%
* Relative/absolute contraindication to DAPT for 12 months (including planned surgeries that cannot be delayed, or subject indicated for chronic oral anticoagulant treatment)
* Calculated creatinine clearance <30 mL/min per Cockcroft-Gault equation (<40mL/min for subjects participating in angiographic follow-up sub-study)
* Hemoglobin <10g/dL
* Platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* White blood cell (WBC) count <3,000 cells/mm3
* Clinically significant liver disease
* Active peptic ulcer/active bleeding from any site
* Bleeding from any site within prior 8 wks requiring active medical/surgical attention
* If femoral access is planned, significant peripheral arterial disease that precludes safe insertion of 6F sheath
* History of bleeding diathesis/coagulopathy/will refuse blood transfusions
* Cerebrovascular accident/transient ischemic attack within past 6 months, or any permanent neurologic defect attributed to CVA
* Known allergy to study stent components, BioNIR or Resolute
* Known allergy to protocol-required concomitant medications: aspirin/DAPT (clopidogrel, prasugrel, ticagrelor)/heparin and bivalirudin/iodinated contrast that cannot be adequately pre-medicated
* Any co-morbid condition that may cause non-compliance with protocol (e.g. dementia, substance abuse) /reduced life expectancy to <24 months (e.g. cancer, severe heart failure, severe lung disease)
* Patient participating/plans to participate in another investigational drug/device clinical trial that has not reached its primary endpoint
* Pregnant/breastfeeding women (women of child-bearing potential must have a negative pregnancy test within 1 wk before treatment)
* Women who intend to become pregnant within 12 months after baseline procedure (sexually active women of child-bearing potential must agree to use a reliable method of contraception from time of screening through 12 months post baseline procedure)
* Patient has received/is on a waiting list for an organ transplant
* Patient receiving/scheduled to receive chemotherapy within 30 days before/any time after the baseline procedure
* Patient receiving oral/intravenous immunosuppressive therapy or has known life-limiting immunosuppressive/autoimmune disease (e.g. HIV); corticosteroids are allowed
* More than 100mm length of planned stenting in the entire coronary tree
* Unprotected left main lesions ≥30%, or planned left main intervention
* Ostial LAD/LCX lesions (stenting of any diseased segment within 5mm of the unprotected left main coronary artery)
* Bifurcation lesions with planned dual stent implantation
* Stenting of lesions due to DES restenosis
* Another lesion in a target/non-target vessel (including all side branches) is present that requires/has high probability of requiring PCI within 12 months after baseline procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1919 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08-28 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Piedmont Healthcare, Atlanta, Georgia, United States
- ZNA Middelheim, Antwerp, Belgium
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada
- Hadassah Hebrew University Medical Center, Jerusalem, Israel
- San Raffaele Hospital, Milan, Italy
- Maasstad Ziekenhuis, Rotterdam, Netherlands
- PAKS, II Oddzial Kardiologiczny, Bielsko-Biala, Poland
- Hospital Meixoeiro, Pontevedra, VIGO, Spain

REFERENCES:
- [Derived] Kandzari DE, Smits PC, Love MP, Ben-Yehuda O, Banai S, Robinson SD, Jonas M, Kornowski R, Bagur R, Iniguez A, Danenberg H, Feldman R, Jauhar R, Chandna H, Parikh M, Perlman GY, Balcells M, Markham P, Ozan MO, Genereux P, Edelman ER, Leon MB, Stone GW. Randomized Comparison of Ridaforolimus- and Zotarolimus-Eluting Coronary Stents in Patients With Coronary Artery Disease: Primary Results From the BIONICS Trial (BioNIR Ridaforolimus-Eluting Coronary Stent System in Coronary Stenosis). Circulation. 2017 Oct 3;136(14):1304-1314. doi: 10.1161/CIRCULATIONAHA.117.028885. Epub 2017 Aug 9. PMID 28794001

RESULTS

PARTICIPANT FLOW:
Groups:
- BioNIR: The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0
  The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
  BioNIR: drug-eluting stent
- Resolute: The Endeavor Resolute Zotarolimus-Eluting Stent System consists of four subsystems:
  1. Endeavor Resolute Stent- a pre-mounted cobalt alloy based stent
  2. Delivery system (Rapid Exchange [RX] Coronary System)
  3. Polymer system
  4. Zotarolimus - drug The Resolute has a nominal drug dose of 1.6µg Zotarolimus per mm2 of the stent surface area.
  Resolute: drug-eluting stent
Period: Overall Study
Arm/Group | BioNIR | Resolute
Started | 958 | 961
Completed | 884 | 878
Not Completed | 74 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioNIR | Resolute | Total
Number analyzed (Participants) | 958 | 961 | 1919
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 509 | 506 | 1015
  >=65 years | 449 | 455 | 904
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.2) | 63.1 (10.3) | 63.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 174 | 382
  Male | 750 | 787 | 1537
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 24 | 25 | 49
  White | 914 | 922 | 1836
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure (TLF)
Description: The primary endpoint of TLF at 12 months was defined as the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of TLF
Groups:
- BioNIR: Participants received The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0
  The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
- Resolute: Participants received The Endeavor Resolute Zotarolimus-Eluting Stent System consists of four subsystems:
  1. Endeavor Resolute Stent- a pre-mounted cobalt alloy based stent
  2. Delivery system (Rapid Exchange [RX] Coronary System)
  3. Polymer system
  4. Zotarolimus - drug The Resolute has a nominal drug dose of 1.6µg Zotarolimus per mm2 of the stent surface area.
Arm/Group | BioNIR | Resolute
Number analyzed (Participants) | 926 | 930
percentage of TLF | 5.4 [4.0 to 7.1] | 5.4 [4.0 to 7.0]

2. Secondary Outcome: Device Success
Description: Clinical: Acute secondary endpoint determined at time of baseline procedure
Time Frame: Determined at time of baseline procedure
Reporting Status: Not Posted

3. Secondary Outcome: TLF
Description: Clinical secondary endpoint to be evaluated at 30 days, 6 months, and 2, 3, 4 and 5 years, defined as the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Major Adverse Cardiac Events
Description: Clinical: MACE; the composite rate of cardiac death, any MI or ischemia-driven TLR
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Target Vessel Failure
Description: Clinical: TVF; the composite rate of death, target vessel related MI or ischemia-driven TVR
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

6. Secondary Outcome: All Cause Mortality
Description: Clinical: The number of patients who die from all causes
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Cardiac Death
Description: Clinical: The number of patients who die of cardiac-related causes
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

8. Secondary Outcome: Myocardial Infarction
Description: Clinical: The number of patients who suffer a myocardial infarction.
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Target Vessel Related MI
Description: Clinical: The number of patients who suffer a MI that is related to the target vessel of the procedure.
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Ischemia Driven TLR
Description: Clinical:
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

11. Secondary Outcome: Ischemia Driven TVR
Description: Clinical:
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

12. Secondary Outcome: Stent Thrombosis
Description: Clinical: ARC definite and probable
Time Frame: 30 days, 6 months, and 1, 2, 3, 4 and 5 years
Reporting Status: Not Posted

13. Secondary Outcome: Angiographic Sub-Study: In-stent and In-segment Late Loss
Description: Secondary Endpoint for angiographic in-stent and in-segment late loss
Time Frame: 13 months
Reporting Status: Not Posted

14. Secondary Outcome: IVUS Sub-Study: In-stent Percent Neointimal Hyperplasia
Description: IVUS: In-stent percent neointimal hyperplasia
Time Frame: 13 months
Reporting Status: Not Posted

15. Secondary Outcome: IVUS Sub-Study: Stent Mal-apposition
Description: IVUS Sub-Study: Stent mal-apposition
Time Frame: 13 months
Reporting Status: Not Posted

16. Secondary Outcome: Lesion Success
Description: Measures whether the lesion was successfully treated.
Time Frame: Determined at time of baseline procedure
Reporting Status: Not Posted

17. Secondary Outcome: Procedure Success
Description: Acute clinical endpoint: The success of the procedure as determined at time of baseline procedure
Time Frame: Determined at time of baseline procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The Investigator monitored the occurrence of adverse events for each subject during the whole course of the trial - baseline and post procedure, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years visits.
Groups:
- BioNIR: Subjects received The BioNIR Ridaforolimus Eluting Coronary Stent System is a single use device/drug combination product comprising:
  * Stent - a mounted Cobalt Chromium (CoCr) alloy based stent
  * Delivery System - Rapid Exchange (RX) Coronary System
  * Polymer matrix coating - Poly n-butyl methacrylate (PBMA) and CarboSil®
  * Ridaforolimus drug - CAS Registry Number: 572924-54-0
  The drug Ridaforolimus is utilized on the stent system at a dose of 1.1 μg/mm2 (with a drug load of 100 μg per 2.75/3.00 x 17 mm stent).
  BioNIR: drug-eluting stent
- Resolute: Subjects received The Endeavor Resolute Zotarolimus-Eluting Stent System consists of four subsystems:
  1. Endeavor Resolute Stent- a pre-mounted cobalt alloy based stent
  2. Delivery system (Rapid Exchange [RX] Coronary System)
  3. Polymer system
  4. Zotarolimus - drug The Resolute has a nominal drug dose of 1.6µg Zotarolimus per mm2 of the stent surface area.
  Resolute: drug-eluting stent
Arm/Group | BioNIR | Resolute
All-Cause Mortality (participants affected / at risk) | 5/958 | 2/961
Serious Adverse Events (participants affected / at risk) | 247/945 | 242/954
Other Adverse Events (participants affected / at risk) | 370/945 | 364/954
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioNIR (N=945) | Resolute (N=954)
blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 1
cardiac disorders (Cardiac disorders) | 159 | 124
ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 3
eye disorderd (Eye disorders) | 1 | 0
gastrointestineal disorders (Gastrointestinal disorders) | 26 | 22
general disorders and administration site condition (General disorders) | 57 | 71
hepatobiliary disorders (Hepatobiliary disorders) | 4 | 2
immune system disorders (Immune system disorders) | 2 | 1
infections and infestations (Infections and infestations) | 15 | 19
injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 | 14
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 1
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 | 4
neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 19
nervous system disorders (Nervous system disorders) | 26 | 27
psychiatric disorders (Psychiatric disorders) | 4 | 0
renal and urinary disorders (Renal and urinary disorders) | 11 | 12
reproductive system and breast disorders (Reproductive system and breast disorders) | 2 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 8 | 16
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures (Surgical and medical procedures) | 3 | 4
Vascular disorders (Vascular disorders) | 8 | 18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BioNIR (N=945) | Resolute (N=954)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 1
Cardiac Disorders (Cardiac disorders) | 159 | 124
ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 3
Eye disorders (Eye disorders) | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 26 | 22
General disorders and administration site conditions (General disorders) | 57 | 71
hepatobiliary disorders (Hepatobiliary disorders) | 4 | 2
immune system disorders (Immune system disorders) | 2 | 1
infections and infestations (Infections and infestations) | 15 | 19
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 | 14
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 1
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 | 4
neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 19
nervous system disorders (Nervous system disorders) | 26 | 27
psychiatric disorders (Psychiatric disorders) | 34 | 0
renal and urinary disorders (Renal and urinary disorders) | 11 | 12
reproductive system and breast disorders (Reproductive system and breast disorders) | 8 | 16
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 8 | 16
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures (Surgical and medical procedures) | 3 | 4
Vascular disorders (Vascular disorders) | 8 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No